CLINICAL TRIAL: NCT03909477
Title: Longitudinal Study of Xenon-129 MRI Imaging of Effects of Cannabis Smoking on Lung Structure and Function
Brief Title: Longitudinal Study of Xenon-129 MRI Imaging Effects of Cannabis Smoking
Status: Recruiting | Type: Observational
Sponsor: Western University, Canada (Other)
Responsible Party: Sponsor
Other Study IDs: ROB0043
Record Dates: First submitted 2019-03-25; First posted 2019-04-10 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Cannabis Use; Cannabis Smoking; Marijuana Smoking; Marijuana Usage
MeSH Terms: conditions — Marijuana Smoking | interventions — Tomography, X-Ray Computed; Respiratory Function Tests; Walk Test; Exercise Test; Hematologic Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Cannabis Smoker: Participants in this group will be current or former cannabis smokers
  Interventions: Diagnostic Test: Hyperpolarized Xenon-129 MRI of the lungs; Diagnostic Test: Computed Tomography (CT); Diagnostic Test: Pulmonary Function Tests (PFTs); Diagnostic Test: Six Minute Walk Test (6MWT); Diagnostic Test: Cardiopulmonary exercise testing (CPET); Diagnostic Test: Sputum analysis; Diagnostic Test: Blood analysis

INTERVENTIONS:
Diagnostic Test: Hyperpolarized Xenon-129 MRI of the lungs — Participants will be imaged using MRI using hyperpolarized xenon-129 gas as a contrast gas
Diagnostic Test: Computed Tomography (CT) — Participants will undergo a CT scan of the thoracic cavity
  Other Names: CT
Diagnostic Test: Pulmonary Function Tests (PFTs) — Participants will have their lung function evaluated using PFTs
  Other Names: PFTs
Diagnostic Test: Six Minute Walk Test (6MWT) — Participants >35 years of age will perform the six minute walk test as a measure of exercise capacity
  Other Names: 6MWT
Diagnostic Test: Cardiopulmonary exercise testing (CPET) — Participants <35 will perform cardiopulmonary exercise testing as a measure of exercise capacity
  Other Names: CPET
Diagnostic Test: Sputum analysis — Participants will provide a sputum sample that will be analysed for eosinophils
Diagnostic Test: Blood analysis — Participants will have their blood drawn and analysed for eosinophil count.

SUMMARY:
This is a longitudinal study of the long-term health impact of cannabis smoking on the lungs. Participants will be followed over a period of 3 years, and impacts of cannabis smoking on the lungs will be measured with magnetic resonance imaging (MRI) using hyperpolarized xenon-129 gas, pulmonary function tests, exercise capacity, computed tomography images and questionnaires.

DETAILED DESCRIPTION:
This is a longitudinal study of the long-term lung health impact of cannabis smoking in adults using xenon-129 (129Xe) MRI over three years.

Males and females between the ages of 18 to 85 years with a history of cannabis smoking will be screened, and those who satisfy all inclusion and exclusion criteria will undergo study visits for up to 3 years, with visits every 12 ± 3 months, for a total of up to four study visits. Each study visit will include collection of patient smoking history and vital signs. At Visit 1 and 4, 129-Xe MRI, spirometry, plethysmography for airways resistance (Raw) and lung volumes, forced oscillation technique (FOT) and multiple breath nitrogen washout (MBNW) for the lung clearance index (LCI) will all be performed pre- and post-bronchodilator. Blood will be drawn for blood eosinophil count, and sputum induction will be done to measure sputum eosinophils. A CT will also be done at Robarts Research Institute, or at University Hospital, London Health Sciences Centre next door to Robarts. Visit 2 will be a telephone call to complete questionnaires. Visit 3 will include spirometry and questionnaires only. Participants 35 years of age or older will complete a six minute walk test (6MWT) for the distance walked (6MWD), pre and post oxygen saturation, perceived dyspnea (Modified Borg Scale) and perceived exertion (Borg's rating of perceived exertion). These participants will complete the St. George's Respiratory Questionnaire (SGRQ).

Participants under the age of 35 will complete Cardio Pulmonary Exercise Testing to assess exercise capacity, and the American Thoracic Society Questionnaire (ATSQ).

ELIGIBILITY:
Inclusion Criteria:

* Patient understands study procedures and is willing to participate in the study as indicated by the patient's signature
* Provision of written, informed consent prior to any study specific procedures
* Males and females aged 18-85
* Current or former cannabis smoker (medicinal or recreational) with or without concurrent tobacco smoking history
* Participant is able to perform reproducible pulmonary function testing (i.e. the 3 best acceptable spirograms have Forced Expiratory Volume in 1 second (FEV1) values that do not vary more than 150 millilitres)
* Participant is able to perform a breathhold for 16s
* FEV1 > 25% predicted
* Forced Vital Capacity (FVC) > 25% predicted and >0.5 litres

Exclusion Criteria:

* Participant is, in the opinion of the investigator, mentally or legally incapacitated, preventing informed consent from being obtained, or cannot read or understand written material
* Participant is medically unstable in the opinion of the Principal Investigator
* Participant has a daytime room air oxygen saturation <90% while lying supine
* Participant is unable to perform spirometry or plethysmography maneuvers
* Patient is pregnant at time of enrolment
* In the opinion of the investigator, patient suffers from any physical, psychological or other condition(s) that might prevent performance of the MRI, such as severe claustrophobia
* Patient has implanted mechanically, electrically or magnetically activated device or any metal in their body, which cannot be removed, including but not limited to pacemakers, neurostimulators, biostimulators, implanted insulin pumps, aneurysm clips, bioprosthesis, artificial limb, metallic fragment or foreign body, shunt, surgical staples (including clips or metallic sutures and/or ear implants) - at the discretion of the MRI Technologist.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Current and former smokers of cannabis
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2030-12-01 (Estimated); Study Completion 2030-12-01 (Estimated)

PRIMARY OUTCOMES:
Changes in airways over time | 3 years
  Measured using Xenon-129 (129-Xe) MRI
Changes in parenchyma over time | 3 years
  Measured using Xenon-129 (129-Xe) MRI
Differences in lung ventilation in cannabis smokers compared to never-smokers and tobacco smokers | 3 years
  Measured using 129-Xe MRI
Differences in perfusion in cannabis smokers compared to never-smokers and tobacco smokers | 3 years
  Measured using 129-Xe MRI
Differences in parenchyma integrity in cannabis smokers compared to never-smokers and tobacco smokers | 3 years
  Measured using 129-Xe MRI
Differences in airways between cannabis-only smokers and cannabis and tobacco smokers | 3 years
  Measured using 129-Xe MRI
Differences in parenchyma between cannabis-only smokers and cannabis and tobacco smokers | 3 years
  Measured using 129-Xe MRI
Dose-response of cannabis use to changes in airways over time | 3 years
  Measured using 129-Xe MRI
Dose-response of cannabis use to changes in parenchyma over time | 3 years
  Measured using 129-Xe MRI

CONTACTS AND LOCATIONS:
Overall Officials: Grace E Parraga, PhD, Principal Investigator — Robarts Research Institute, The University of Western Ontario
Locations (1):
- Robarts Research Institute; The University of Western Ontario; London Health Sciences Centre, London, Ontario, Canada